CLINICAL TRIAL: NCT04715334
Title: Effectiveness in Improving Gait and Feasibility of a Transcutaneous Electrical Stimulation Garment in Children With Cerebral Palsy in Singapore
Brief Title: Can Transcutaneous Electrical Stimulation Garment Improve Gait in Children With Cerebral Palsy?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: KK Women's and Children's Hospital (Other Government)
Collaborators: Inerventions AB (Unknown)
Responsible Party: Principal Investigator, Ng Zhi Min, Senior Consultant, KK Women's and Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020/2150
Record Dates: First submitted 2020-12-07; First posted 2021-01-20 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Cerebral Palsy; Spasticity, Muscle
Keywords: gait; electrical stimulation
MeSH Terms: conditions — Cerebral Palsy; Muscle Spasticity

STUDY DESIGN:
Intervention Model Description: pre and post intervention comparison
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm study (Experimental): The intervention is the Mollii suit which is fitted and programmed by the Mollii suit distributor, Inerventions and will be administered by trained physiotherapists from KKH. Participants will be involved in the Intervention phase of the study for 4 weeks with treatment duration of 60 min/ session every day.
  Interventions: Device: Mollii suit

INTERVENTIONS:
Device: Mollii suit — The Mollii suit is a new technology of electrical stimulation in the form of whole-body garment with multiple electrodes individually programmed to stimulate the selected muscles. Based on preliminary studies, it is suggested that the Mollii suit improves spasticity. Recent studies also proposed that it improves mobility, gait, function and quality of life. However, these studies are based on qualitative and subjective measures.

SUMMARY:
Living with cerebral palsy is challenging for the child as well as the family charged with their care and support needs. Many families seek effective and sustainable interventions to improve gait of their children with cerebral palsy. The Mollii suit is a non-invasive therapeutic technology using electrical stimulation in the form of whole-body garment with multiple electrodes individually programmed to stimulate selected muscles. This study aims to examine if the Mollii suit improve gait in ambulant children with cerebral palsy and if the Mollii suit is acceptable and tolerable to children with cerebral palsy. We will recruit up to 20 children with cerebral palsy. This study will evaluate change in gait and function following a four-week intervention period using a protocol of wearing the Mollii suit at home for one hour every day for four weeks using instrumented 3-dimensional gait analysis and objective standardised assessment tools.

DETAILED DESCRIPTION:
BACKGROUND

Living with cerebral palsy is challenging for the child as well as the family charged with their care and support needs. Many families seek effective and sustainable interventions to improve gait of their children with cerebral palsy. An intervention that could be used in the home setting, assessed periodically by health care professionals of a tertiary pediatric centre, that has a benefit on gait and motor function in children with cerebral palsy might be feasible to families in the local Singapore healthcare setting. The Mollii suit is a non-invasive therapeutic technology using electrical stimulation in the form of whole-body garment with multiple electrodes individually programmed to stimulate selected muscles. Based on small preliminary studies, it is suggested that the Mollii suit improves mobility, gait, function and quality of life.

OBJECTIVES

This study aims to examine the effectiveness of the Mollii suit in improving gait in children with cerebral palsy. It also aims to determine the value of the Mollii suit by evaluating the acceptability, tolerance and compliance of the Mollii suit in children with cerebral palsy.

METHODOLOGY

This is a single-centre study that will recruit up to 20 children with cerebral palsy, GMFCS I-III. This study will evaluate change in gait and function following a four-week intervention period using a protocol of wearing the Mollii suit at home for one hour every day for four weeks using instrumented 3-dimensional gait analysis and objective standardised assessment tools. Primary outcome is improvement in gait, measured using the Gait Profile Score, Gait Deviation index, gait speed and cadence. Secondary outcomes include changes in functional assessments such as Functional Assessment Questionnaire (FAQ), Gross Motor Function Measure (GMFM), 10 metre walk test, Goal attainment Scale (GAS) and quality of life measures.

ELIGIBILITY:
Inclusion Criteria:

* Aged 4-18
* GMFCS level I to III
* Spasticity as the dominant motor feature
* Children agree to wear the Mollii suit as per procedures and consent to the study
* Parents/carers agree to assist their child to wear the Mollii suit as per procedures
* Medical practitioner's approval

Exclusion Criteria:

* Individuals with electrical implanted stimulatory device
* Individuals with medical devices that are affected by magnets, such as programmable shunts.
* Individuals with cardiovascular diseases, infectious diseases, malignance (cancer), fever, pregnancy, rashes or skin problems.
* Individuals who have had Botulinum toxin done 6 months prior intervention or soft tissue release surgery done 6 months prior intervention.
* Individuals who have had change in oral medication for spasticity 1 month prior intervention.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-12-08 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Gait Profile Score (GPS) | 1 month post intervention
  GPS is a single index measure that summarises the overall deviation of kinematic gait data relative to normative data. It ranges from 0 to 30, the higher the score, the more severe the gait. We will measure change in GPS pre and post intervention.
Change in Gait Profile Score (GPS) | 2 months post intervention
  GPS is a single index measure that summarises the overall deviation of kinematic gait data relative to normative data. It ranges from 0 to 30, the higher the score, the more severe the gait. We will measure change in GPS pre and post intervention.
Change in Gait deviation index (GDI) | 1 month post intervention
  GDI provides a numerical value that expresses overall gait pathology (ranging from 0 to 100, where 100 indicates the absence of gait pathology). The higher the GDI, the better the result.
Change in Gait deviation index (GDI) | 2 months post intervention
  GDI provides a numerical value that expresses overall gait pathology (ranging from 0 to 100, where 100 indicates the absence of gait pathology). The higher the GDI, the better the result.
Change in Gait speed (metre/sec) | 1 month post intervention
  The faster the gait speed, the better the result.
Change in Gait speed (metre/sec) | 2 months post intervention
  The faster the gait speed, the better the result.
Change in Cadence (steps/ minute) | 1 month post intervention
  The higher the cadence, the better the result.
Change in Cadence (steps/ minute) | 2 months post intervention
  The higher the cadence, the better the result.

SECONDARY OUTCOMES:
Change in Gross motor function measure (GMFM) | 1 month post intervention
  GMFM is an assessment tool designed and evaluated to measure changes in gross motor function with intervention in children with cerebral palsy. The closer the score to 100%, the better the score.
Change in Gross motor function measure (GMFM) | 2 months post intervention
  GMFM is an assessment tool designed and evaluated to measure changes in gross motor function with intervention in children with cerebral palsy. The closer the score to 100%, the better the score.
Change in Functional Assessment Questionnaire (FAQ) | 1 month post intervention
  FAQ is a 10 point scale (with 10 being most able) which was designed specifically to be used as an outcome measure in individuals with physical disability. The higher the score the better the result.
Change in Functional Assessment Questionnaire (FAQ) | 2 months post intervention
  FAQ is a 10 point scale (with 10 being most able) which was designed specifically to be used as an outcome measure in individuals with physical disability. The higher the score the better the result.
Change in EQ5D | 1 month post intervention
  EQ5D is a standardised measure of health status to provide a simple, generic measure of health for clinical and economic appraisal. The descriptive system comprises 5 dimensions. Score ranges from 5 to 15. The higher score the poorer the result. The EQ VAS records the respondent's self-rated health on a vertical, visual analogue scale 0-100. The higher the score, the better the self-rated health.
Change in EQ5D | 2months post intervention
  EQ5D is a standardised measure of health status to provide a simple, generic measure of health for clinical and economic appraisal. The descriptive system comprises 5 dimensions. Score ranges from 5 to 15. The higher score the poorer the result. The EQ VAS records the respondent's self-rated health on a vertical, visual analogue scale 0-100. The higher the score, the better the self-rated health.
Change in ICF-CY ratings | 1 month post intervention
  The WHO International Classification of Functioning, Disability and Health, Children & Youth version (ICF-CY) is a measure to grade function of activities of daily living (ADLs). Few ICF-CY categories have been selected and graded based on the frequency, intrusiveness or severity of the specific impairment. In each category, rating ranges from 0 to 4. The higher the rating, the worse the outcome.
Change in ICF-CY ratings | 2 months post intervention
  The WHO International Classification of Functioning, Disability and Health, Children & Youth version (ICF-CY) is a measure to grade function of activities of daily living (ADLs). Few ICF-CY categories have been selected and graded based on the frequency, intrusiveness or severity of the specific impairment. In each category, rating ranges from 0 to 4. The higher the rating, the worse the outcome.
Compliance | 1 month post intervention
  Compliance is measured using log of use of mollii suit.
Compliance | 2 months post intervention
  Compliance is measured using log of use of mollii suit.
Acceptance | 1 month post intervention
  Acceptance to the mollii suit is evaluated qualitatively using an open-ended questionnaire filled up by patient and caregivers
Acceptance | 2 months post intervention
  Acceptance to the mollii suit is evaluated qualitatively using an open-ended questionnaire filled up by patient and caregivers

CONTACTS AND LOCATIONS:
Overall Officials: Zhi Min Ng, MBBS, Principal Investigator — KK Women's and Children's Hospital
Locations (1):
- KKWCH, Singapore, Singapore

REFERENCES:
- [Background] Mills PB, Dossa F. Transcutaneous Electrical Nerve Stimulation for Management of Limb Spasticity: A Systematic Review. Am J Phys Med Rehabil. 2016 Apr;95(4):309-18. doi: 10.1097/PHM.0000000000000437. PMID 26829077
- [Background] Wright PA, Durham S, Ewins DJ, Swain ID. Neuromuscular electrical stimulation for children with cerebral palsy: a review. Arch Dis Child. 2012 Apr;97(4):364-71. doi: 10.1136/archdischild-2011-300437. PMID 22447997

DOCUMENTS (1):
  • Study Protocol (2020-03-30): https://cdn.clinicaltrials.gov/large-docs/34/NCT04715334/Prot_000.pdf